CLINICAL TRIAL: NCT02463513
Title: RIBOGENE: Optimisation of Riboflavin Status in Hypertensive Adults With a Genetic Predisposition to Elevated Blood Pressure
Acronym: RIBOGENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ulster (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OREC 12/NI/0136
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Participants With the MTHFR 677TT Genotype
Keywords: Riboflavin; Blood pressure; MTHFR; Methylenetetrahydrofolate reductase
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo comparator
- Treatment 2 (Active Comparator)
  Interventions: Dietary Supplement: 1.6mg riboflavin (Vitamin B2)
- Treatment 3 (Active Comparator)
  Interventions: Dietary Supplement: 10mg riboflavin (Vitamin B2)

INTERVENTIONS:
Dietary Supplement: Placebo comparator — 2 week placebo washout + 16 weeks intervention (placebo)
  Arms: Treatment 1
Dietary Supplement: 1.6mg riboflavin (Vitamin B2) — 2 week placebo washout + 16 weeks intervention (1.6mg riboflavin per day)
  Arms: Treatment 2
Dietary Supplement: 10mg riboflavin (Vitamin B2) — 2 week placebo washout + 16 weeks intervention (10mg riboflavin per day)
  Arms: Treatment 3

SUMMARY:
Approximately 10% of the world's population have a particular genetic makeup (known as the TT genotype) that may increase their risk of having higher blood pressure. Previous work conducted by the investigators research group at the University of Ulster, in collaboration with clinical colleagues from across Northern Ireland, in premature CVD patients and hypertensive adults generally has demonstrated that a dietary level of riboflavin (1.6mg/d) decreases blood pressure, specifically in those with the TT genotype. To date, the blood pressure lowering effects of higher doses of riboflavin in individuals with the TT genotype is not known. The aim of this study is to investigate whether supplementation with riboflavin at a low dose supplemental level (10mg/d) can decrease blood pressure more effectively than the dietary level (1.6mg/d) by optimising riboflavin status and normalising MTHFR activity. This aim will be achieved by conducting a double-blind placebo-controlled intervention study over a 16 week period.

Participants will be recruited from cohorts screened for the methylenetetrahydrofolate reductase (MTHFR) C677T polymorphism. Those identified with the TT genotype (homozygous for the polymorphism) that wish to participate in this research will be asked to attend a baseline and week-16 appointment and will be asked to take a daily riboflavin (1.6 or 10mg/d) or placebo capsule for the duration of the study. At each appointment a blood sample will be taken and blood pressure, height, weight and waist circumference will be measured. If the results of this study show that intervention with a higher dose of riboflavin can lower blood pressure more effectively in individuals with the TT genotype this will have important implications for those responsible for the management of blood pressure. The findings will be of particular relevance in populations with a higher prevalence of the polymorphism.

DETAILED DESCRIPTION:
Recruitment - Potential participants will be identified and recruited via GP practices, hospital outpatient clinics, pharmacies and workplaces throughout Northern Ireland. A letter of invitation and a study package containing a participant information sheet to explain the study, a consent form and a buccal swab DNA collection kit will be included.

Inclusion / Exclusion The main inclusion criteria are that individuals must have the TT genotype. Exclusion criteria includes a history of gastrointestinal, hepatic, renal or haematological disorders, B-vitamin supplements consumer (including multi-vitamins containing B-vitamins), anticonvulsant therapy or any other drugs known to interfere with folate/B-vitamin metabolism. Suitable individuals that participated in the screening process will be contacted and invited to participate in the intervention study. Participants will be given at least forty eight hours to consider the written information and decide if they wish to participate.

Study Design

Participants with the TT genotype who have given informed consent will be stratified by blood pressure and subsequently randomised to receive placebo, low dose (1.6mg/d) or low supplemental dose (10mg/d) riboflavin for the 16 week intervention period. It is important to be aware that no upper limit has been established for this water-soluble B-vitamin and there are no safety concerns regarding these doses of riboflavin or indeed higher doses (including 25mg/d) administered in previous studies (Madigan et al. 1998).

Participants, depending on geographical location, will be asked to attend two appointments (Baseline and week 16) at the participants local GP Practice, The Clinical Translational Research and Innovation Centre (CTRIC) at Altnagelvin Area Hospital, The Welcome Trust-Wolfson Northern Ireland Clinical Research Facility (NICRF) Belfast City Hospital, the Northern Ireland Centre for Food & Health (NICHE) (University of Ulster, Coleraine) or at another convenient location. At both sampling points blood pressure (SBP/DBP mmHg) will be measured, a 30ml blood sample will be taken by a trained phlebotomist and the patient's height (m), weight (kg), waist circumference (cm) and BMI (kg/m2) will be measured. A detailed health and lifestyle questionnaire will collect information on medical and family history, medication and supplement use and dietary intake.

Statistical analysis Statisticalanalysis will be performed using SPSS (Statistical Package for Social Sciences, Version 17.0; SPSS UK Ltd, Chersey, United Kingdom). Data that is not normally distributed will be transformed to obtain normality before statistical analysis is performed. Data will then be analysed to investigate if any differences exist in the BP response between the two riboflavin treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old

Exclusion Criteria:

* History of gastrointestinal; Hepatic; Renal or haematological disorders
* Taking B-vitamin supplements (including multi-vitamins containing B-vitamins), anticonvulsant therapy or any other drugs known to interfere with folate/B-vitamin metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 16 weeks
  The aim of this study is to investigate whether a low dose supplemental level (10mg/d) of riboflavin can decrease blood pressure more effectively than the dietary level (1.6mg/d) by optimising riboflavin status and normalising MTHFR activity.

SECONDARY OUTCOMES:
Erythrocyte Glutathione Reductase Activation Coefficient (EGRAC) | 16 weeks
  Indicator of Vitamin B2 status
Plasma Homocysteine | 16 weeks
Red cell folate | 16 weeks
Vitamin B12 | 16 weeks
Vitamin B6 | 16 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Northern Ireland Clinical Research Facility (NICRF), Belfast, N.Ireland
  - Human Intervention Studies Unit, University of Ulster, Coleraine, N.Ireland
  - Clinical Translational Research and Innovation Centre (C-TRIC), Londonderry, N.Ireland